CLINICAL TRIAL: NCT07355478
Title: Asia Myelodysplastic Syndrome (MDS) Registry
Status: Not yet recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA056-1131
Record Dates: First submitted 2025-11-28; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Myelodysplastic Syndromes (MDS)
Keywords: Myelodysplastic syndromes (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Group 1: Participants diagnosed with myelodysplastic syndromes (MDS)
  Interventions: Drug: Prescribed treatments for myelodysplastic syndromes (MDS)

INTERVENTIONS:
Drug: Prescribed treatments for myelodysplastic syndromes (MDS) — According to the product label

SUMMARY:
The purpose of this study is to provide a contemporary view and offer invaluable insights into the demographic profiles, clinical characteristics, treatments, and real-world outcomes of individuals with myelodysplastic syndromes (MDS) in Asia.

ELIGIBILITY:
Inclusion Criteria:

Retrospective enrolment of Myelodysplastic Syndrome (MDS) participants:

* Aged at least 18 years at initial diagnosis of MDS
* Diagnosed with MDS according to World Health Organization (WHO) 2008, WHO 2016, or WHO 2022 criteria between 1 January 2019 and 31 December 2022; and
* Diagnosed with MDS within 100 days from the date of diagnostic bone marrow (BM) aspirate

Inclusion criteria for the prospective enrolment of MDS participants:

* Aged at least 18 years at initial diagnosis of MDS; and
* Diagnosed with MDS according to World Health Organization (WHO) 2008, WHO 2016, or WHO 2022 criteria between 1 October 2025 and 30 September 2026; and
* Diagnosed with MDS within 100 days from the date of diagnostic BM aspirate

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry will include adults who were/are newly diagnosed with myelodysplastic syndromes (MDS) in Asia (Singapore, South Korea and Taiwan).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-01-28 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Participant age | Baseline
Participant sex | Baseline
Participant race | Baseline
Participant weight | Baseline
Participant height | Baseline
Participant body mass index (BMI) | Baseline
Participant smoking status | Baseline
Participant drinking status | Baseline
Family history of MDS or other hematopoietic cancers | Baseline
Participant myelodysplastic syndromes diagnosis information | Baseline
Participant Eastern Cooperative Oncology Group (ECOG) Performance status at diagnosis | Baseline
Participant comorbidities at diagnosis | Baseline
Participant Charlson comorbidity index (CCI) score at diagnosis | Baseline
Prior clinical diagnosis of other cancers | Baseline
Prior clinical diagnosis of hematological diseases | Baseline
Anemia status at diagnosis | Bseline
Thrombocytopenia status at diagnosis | Baseline
Neutropenia status at diagnosis | Baseline
Iron overload status at diagnosis | Baseline
Red blood cell (RBC) transfusion dependence status at diagnosis | Baseline
International Prognostic Scoring System (IPSS) score at diagnosis | Baseline
Revised International Prognostic Scoring System (IPSS-R) score at diagnosis | Baseline
Molecular International Prognostic Scoring System (IPSS-M) score at diagnosis | Baseline
Bone marrow aspirate results | Baseline and up to 2-years
Presence of dysplasia | Baseline and up to 2-years
Cytogenetic test results | Baseline and up to 2-years
Mutation test results at diagnosis | Baseline
Complete blood count test results at diagnosis | Baseline
Mean corpuscular volume (MCV) | Baseline and up to 2-years
C-reactive protein (CRP) | Baseline and up to 2-years
Serum ferritin (SF) level | Baseline and up to 2-years
Serum erythropoietin levels | Baseline and up to 2-years
Lactate dehydrogenase (LDH) | Baseline and up to 2-years

SECONDARY OUTCOMES:
Initial treatment received following diagnosis | Baseline
Prior treatments and concomitant medications received | Baseline
Subsequent treatments received | Up to 2-years
Time from diagnosis to treatment initiation | Baseline
Treatment duration | Up to 2-years
Real-world overall survival (rwOS) | Baseline and up to 2-years
Time to disease-risk progression (per IPSS-R) | Baseline and up to 2-years
Time to acute myeloid leukemia (AML) progression | Baseline and up to 2-years
Time to iron overload | Baseline and up to 2-years
Overall response rate (ORR) | Baseline and up to 2-years
Duration of response (DOR) | Baseline and up to 2-years
Real-world relapse-free survival (rwRFS) | Baseline and up to 2-years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Seoul National University Hospital, Seoul, South Korea
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts